CLINICAL TRIAL: NCT01966380
Title: An Open Randomised, Prospective, Crossover, Proof of Concept (Design Validation) Clinical Investigation to Caompare the Performance and Safety of Wound Dressing(Leia) Compared to and Hydroactive Surgical Dressing on Low to Highly Exuding Wounds
Brief Title: Proof of Concept (Design Validation) in Patient With Hard to Heal Wounds Such as Pressure Ulcer, Diabetic Foot Ulcer and Leg Ulcer, Leia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Leia
Record Dates: First submitted 2013-10-09; First posted 2013-10-21 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Leg Ulcer; Diabetic Foot Ulcer; Pressure Ulcer
MeSH Terms: conditions — Leg Ulcer; Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device, dressing (Experimental): Intervention: Device, Leia dressing
  Interventions: Device: Leia
- Dressing , device (Active Comparator): Intervention: Device: Hydroactive surgical dressing
  Interventions: Device: Leia

INTERVENTIONS:
Device: Leia
  Other Names: Leia consist of conducting and absorbing part.; Device: Hydroactive surgical dressing; It is a synergetic combination of a hydroactive surgical dressing

SUMMARY:
The purpose of this reseach study is to determine Mölnlycke Health Care´s Leia dressing performance properties is fulfilled and that the dressing is safe when used on wound types such as pressure ulcer, leg ulcer, and diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Low to highly exuding chronic wound(wound history > 2 months) such as Leg Ulcer, Pressure Ulcer Category III to IV or Diabetic Foot Ulcer
* Male of female, 18 years and above
* Signed Informed Consent Form

Exclusion Criteria:

* Pregnancy or lactation
* Wound size not suitable for the wound dressing size
* Known allergy/hypersensitivity to any of the components in the dressing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska clinical trial center, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Cross-over Assignment Leia: First intervention Leia, 5 Days, then second intervention Hydroactive surgical dressing 5 Days.
- Cross-over Assignment Hydroactive Surgical Dressing: First intervention Hydroactive surgical dressing 5 Days, then second intervention Leia, 5 Days..
Period: Overall Study
Arm/Group | Cross-over Assignment Leia | Cross-over Assignment Hydroactive Surgical Dressing
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Leia and Hydroactive Surgical Dressing: In the case of this study, participants served as their own control.
Arm/Group | Leia and Hydroactive Surgical Dressing
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 71 [59 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  Sweden | 6

OUTCOME MEASURES:

1. Primary Outcome: Absorption of Wound Exudates.
Description: Absorption capacity measured subjectively: NA/POOR/GOOD/VERY GOOD/EXCELLENT
Time Frame: 2-3 weeks
Population: Participants served as their own controll, those the total amount of participants is reflekted in both of the outcome measurements.
Measure: Number; unit: Total no. assess. in each wounddressing
Units Other Than Participants: Abosorbtion capacity of wounddressing
Groups:
- Leia: Intervention: Device, Leia dressing Cross-over design, the patient was his own controll. 6 patients were treated in total.
- Hydroactivate Surgical Dressing: Intervention: Device, Hydroactivate surgical dressing. Cross-over design, the patient was his own controll. 6 patients were treated in total.
Arm/Group | Leia | Hydroactivate Surgical Dressing
Number analyzed (Participants) | 6 | 6
Number analyzed (Abosorbtion capacity of wounddressing) | 20 | 21
Total no. assess. in each wounddressing
  Good | 8 | 7
  Very good | 5 | 5
  Excellent | 0 | 1
  NA | 7 | 8
  Poor | 0 | 0

ADVERSE EVENTS:
Groups:
- Hydroactive Surgical Dressing: Intervention: Device: Hydroactive surgical dressing
  Cross-over design, the patient was his own controll. 6 patients were treated in total.
Arm/Group | Leia | Hydroactive Surgical Dressing
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leia (N=6) | Hydroactive Surgical Dressing (N=6)
additional wound (Skin and subcutaneous tissue disorders) | 3 | 0 — Additional wound outside target wound

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other